CLINICAL TRIAL: NCT02675062
Title: The Effect of Total Knee Arthroplasty on Habitual Physical Activity, Sedentary Behaviour and Health Outcomes in Patients With Osteoarthritis
Brief Title: Habitual Physical Activity and Sedentary Behavior Following Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Rebecca Meiring, Dr, University of Witwatersrand, South Africa
Other Study IDs: M150323
Record Dates: First submitted 2016-01-29; First posted 2016-02-05 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Knee Osteoarthritis
Keywords: Accelerometry; Osteoarthritis; Habitual physical activity; Sedentary behaviour; Knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether habitual physical activity and sedentary behaviour improve six weeks and between three to six months after total knee replacement surgery in people with osteoarthritis.

DETAILED DESCRIPTION:
The aims of this study are to

1. describe habitual physical activity and sedentary behaviour patterns in knee osteoarthritis patients who are scheduled for total knee arthroplasty,
2. investigate the effects of unilateral primary total knee arthroplasty on objectively and subjectively measured physical activity, sedentary behaviour and health outcomes of knee OA patients and
3. compare subjective measures of functional ability and sedentary behaviour (questionnaires) with objective measures of habitual physical activity and sedentary behaviour (accelerometry) both before and after total knee arthroplasty.

Study design:

This a longitudinal follow-up study of a cohort of participants who have been diagnosed with knee osteoarthritis and who will all be undergoing total knee arthroplasty. After enrolment into the study, baseline assessments will be done prior to total knee arthroplasty. After total knee arthroplasty, participants will be followed-up and the same assessments done at baseline will also be done at 6 weeks, and 3 to 6 months post-operatively. Habitual physical activity and sedentary behaviour will be measured using accelerometry (Actigraph GTX3+ and ActivPal monitors) at the specific time points.The ActiGraph will be worn by participants for 24 hours/day for seven days at each of the assessment time points. It will be attached to an elastic nylon strap which the participants can wear as a belt around the waist on the side of right/left hip (depending on which knee is being operated on). Thus, the ActiGraph will be worn on the side of left hip if the total knee arthroplasty is on the left knee and vice versa. Participants will be asked to remove the ActiGraph when showering, bathing or swimming. After seven days of accelerometer wear, the accelerometers will be collected at the next possible visit to the hospital or arrangement will be made for collection from participants at a location most convenient to them. An ActivPAL will be taped to the thigh of the patient with waterproof taping and the patient will be asked to keep the ActivPAL on for the same amount of time as the ActiGraph. The ActivPAL can be covered with waterproof taping therefore, there will be no need to remove the ActivPAL when showering, bathing or swimming. The ActivPAL will be collected at the same time as the ActiGraph. In addition, general health, functional ability, generic quality of life and sleep and pain questionnaires will be conducted at each time point on each participant.

Study Site:

The study will be conducted at the Charlotte Maxeke Academic Hospital in Johannesburg, South Africa. It is an accredited central hospital with about 1088 beds serving patients from across Gauteng and neighbouring provinces. The hospital is situated in Parktown and also, serves as the main teaching hospital for the University of the Witwatersrand, Faculty of Health Sciences. Study participants will be recruited from the Division of Orthopaedics in the hospital. This hospital is chosen because: (1) it is a tertiary hospital that runs several specialist clinics including the Orthopaedic Division where total knee arthroplasty is performed and (2) there is a collaboration between the Academic staff of the Faculty of Health Sciences of University of the Witwatersrand and the hospital Staff for teaching and research which will facilitate accessibility to patients.

Sample Size Determination:

Based on an anticipated 2% decrease in the amount of time spent in sedentary behaviour per day (which, for an average 16 hour day, equates to a 20 minute reduction), a sample size calculation shows that a total sample of 107 participants will be required in this study to detect a significant effect of knee arthroplasty on sedentary behaviour with a power of 80%.

The effect of the total knee arthroplasty on the change in habitual physical activity and sedentary behaviour will be assessed between the three timepoints (baseline, six weeks and three to six months).

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of knee osteoarthritis
* Kellgren and Lawrence grade 4 severity of knee osteoarthritis
* refractory to analgesics for at least six months
* undergoing primary or first-time single total knee arthroplasty
* are ambulant with or without assistive devices

Exclusion Criteria:

* use assistive ambulatory devices for mobility problems other than knee osteoarthritis
* scheduled for bilateral knee arthroplasty, a second knee arthroplasty or revision
* scheduled for total hip replacement
* co-morbidities or medical conditions that affect physical activity such as congestive heart failure, stroke and other neurological problems, chronic obstructive pulmonary disease, gout and/or sepsis
* rheumatoid arthritis
* undergoing another surgery following the knee arthroplasty
* non-ambulant or wheel chair-bound

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all knee osteoarthritis patients receiving care at the Charlotte Maxeke Johannesburg Academic Hospital. Patients will be recruited from the Orthopaedic Division of the hospital. The participants for this study will be knee osteoarthritis patients scheduled (on surgical waiting list) for a single primary total knee arthroplasty. Knee osteoarthritis will be diagnosed based on clinical criteria as defined by the American Rheumatism Association. The grade of knee osteoarthritis will be graded using the Kellgren and Lawrence classification of severity.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-08; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Habitual physical activity level | Baseline
  Measured using the ActiGraph accelerometer
Habitual physical activity level | Six weeks post-op
  Measured using the ActiGraph accelerometer
Habitual physical activity level | Between three and six months post-op
  Measured using the ActiGraph accelerometer
Time spent in sedentary behaviour | Baseline
  Measured using the activPAL accelerometer
Time spent in sedentary behaviour | Six weeks post-op
  Measured using the activPAL accelerometer
Time spent in sedentary behaviour | Between three and six months post-op
  Measured using the activPAL accelerometer

SECONDARY OUTCOMES:
Knee osteoarthritis-specific quality of life | Baseline, 6 weeks post-op, between 3 and 6 months post-op
  Measured using Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Activity | Baseline, 6 weeks post-op, between 3 and 6 months post-op
  Measured using the UCLA activity index (self-report)
Pain | Baseline, 6 weeks post-op, between 3 and 6 months post-op
  Measured using a visual analogue scale
Sleep quality | Baseline, 6 weeks post-op, between 3 and 6 months post-op
  Measured using a sleep questionnaire
Total summed score of pain, activity, sport and recreation function and knee-related quality of life. | Baseline, 6 weeks post-op, between 3 and 6 months post-op
  Measured using the Knee injury and Osteoarthritis Outcome Score (KOOS)
Score of pain and physical disability | Baseline, 6 weeks post-op, between 3 and 6 months post-op
  Measured using the Oxford Knee Score (OKS)
Knee functional score | Baseline, 6 weeks post-op, between 3 and 6 months post-op
  Measured using the Knee Society Clinical Rating System (KSS)
Patient functional score | Baseline, 6 weeks post-op, between 3 and 6 months post-op
  Measured using the Knee Society Clinical Rating System (KSS)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Meiring, PhD, Study Director — University of Witwatersrand, South Africa
Locations (1):
- Division of Orthopaedics, Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meiring RM, Frimpong E, Mokete L, Pietrzak J, Van Der Jagt D, Tikly M, McVeigh JA. Rationale, design and protocol of a longitudinal study assessing the effect of total knee arthroplasty on habitual physical activity and sedentary behavior in adults with osteoarthritis. BMC Musculoskelet Disord. 2016 Jul 13;17:281. doi: 10.1186/s12891-016-1141-5. PMID 27411316